CLINICAL TRIAL: NCT01305512
Title: Pharmacokinetic, Safety and Tolerability Study of SPARC1028
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLR_10_28
Record Dates: First submitted 2011-02-24; First posted 2011-02-28 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor in Advanced Stage
Keywords: Solid; Tumor; Taxane
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPARC1028 (Experimental)
  Interventions: Drug: SPARC1028

INTERVENTIONS:
Drug: SPARC1028 — SPARC1028 administration as 30-minute intravenous infusion once a week for 3 weeks, followed by 1 week of rest

SUMMARY:
Evaluation of pharmacokinetic profile of SPARC1028

DETAILED DESCRIPTION:
This is a phase I study of SPARC1028 and recommend phase II dose of SPARC1028 administered once a week for 3 weeks, followed by 1 week of rest.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of solid tumor in advanced stage which taxane-based therapy is a rational treatment option.
* Age ≥18 years
* ECOG Performance Status ≤ 1.
* Estimated life expectancy of at least 12-weeks;

Exclusion Criteria:

* Any malignancy within past 5-years, except non-melanoma skin cancer, cervical intraepithelial neoplasia, or in situ cervical cancer
* Known hypersensitivity to the study drugs
* Treatment with any anti-cancer agents within 28 days of study entry
* Presence of clinically evident active CNS metastases, including leptomeningeal involvement, requiring steroid or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) during dose escalation | One 21-day treatment cycle
  MTD for SPARC1028 will be determined as dose below the dose at which DLT (Dose Limiting Toxicity) is seen for ≥ 2 subjects

SECONDARY OUTCOMES:
Establishing pharmacokinectic profile at each dose level for SPARC1028 | One 21-day treatment cycle
  Plasma levels of SPARC1028 will be determined and PK parameters viz., Cmax, AUC0-t, AUC0-∞, MRT, Tmax, t½, Kel, Vd, Cl for SPARC1028 will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Buffalo, New York, United States